CLINICAL TRIAL: NCT06488781
Title: Antibiotic Prophylaxis to Prevent Obesity-Related Induction Complications in Nulliparae at Term 2.0 (APPOINT 2.0): A Multi-center Randomized Controlled Trial
Brief Title: Antibiotic Prophylaxis to Prevent Obesity-Related Induction Complications in Nulliparae at Term 2.0
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: University of Alabama at Birmingham (Other); University of Florida (Other); Duke University (Other); Case Western Reserve University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: APPOINT 2.0
Record Dates: First submitted 2024-05-28; First posted 2024-07-05 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Obesity in Pregnancy; Labor Complication
MeSH Terms: conditions — Pregnancy in Obesity; Obstetric Labor Complications | interventions — Azithromycin; Cefazolin

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned 1:1 to receive either the prophylactic antibiotic regimen or placebos during labor induction.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study participants, clinical personnel, and members of the research team responsible for collecting clinical outcomes will be blinded to the treatment group allocation. The research pharmacist at each site and the research analyst generating the randomization scheme will be the only study team members to know the treatment group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prophylactic antibiotics (Active Comparator): Azithromycin 500 milligrams intravenously once and cefazolin 2 grams intravenously every 8 hours for up to three doses
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Placebos, similar in appearance, in place of azithromycin and cefazolin
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — Azithromycin 500 milligrams intravenously once and cefazolin 2 grams intravenously every 8 hours for up to three doses
  Other Names: Cefazolin
  Arms: Prophylactic antibiotics
Drug: Placebo — Placebo given in place of other two active drugs
  Arms: Placebo

SUMMARY:
Obesity increases the risk of pregnancy complications, including puerperal infections and cesarean delivery, and risk rises with increasing body mass index (BMI). Since obese women are more likely to have comorbidities that would necessitate delivery prior to their due date (i.e. prior to 40 weeks gestation), and class III obesity specifically is an indication for delivery by 39 weeks, these patients have a high rate of labor induction. In nulliparous women from the general population (obese and non-obese), labor induction at 39 weeks (compared to expectant management) is associated with less maternal morbidity and a lower cesarean rate. Researchers previously conducted a pilot randomized placebo-controlled trial in obese, nulliparous women undergoing labor induction at term and found that the cesarean delivery rate was lower in women who received a prophylactic antibiotic regimen during labor compared with those who received the placebo. Researchers proposed multi-center trial aims to test this hypothesis in a large sample with adequate power to determine whether prophylactic antibiotics during labor are associated with a decrease in the rate of cesarean delivery in term, nulliparous, obese women. If the findings from the pilot trial are confirmed, this would represent a novel intervention to decrease the cesarean delivery rate in a subset of women at highest risk for cesarean-related complications.

DETAILED DESCRIPTION:
This is a multi-center randomized placebo-controlled trial in which nulliparous women with obesity who are undergoing induction of labor at term and not receiving IAP for GBS will be recruited (n=787). The participants will be randomized 1:1 to receive either prophylactic antibiotics during their labor induction (azithromycin 500 milligrams intravenously once and cefazolin 2 grams intravenously every 8 hours for up to three doses) or like-appearing placebos. The participants and their obstetrical providers will be blinded to the study intervention. The study will be conducted with an identical protocol at five study sites. Trained research nurses/assistants at each study site will consent and enroll participants, collect biospecimens, and collect demographic information and data on pregnancy and neonatal outcomes, and will convey this data to the primary site for analysis.

Researchers hypothesize that the group that receives the study drug regimen of prophylactic antibiotics during induction of labor will have a lower rate of cesarean delivery than the group that receives the placebo. They also hypothesize that the group that receives the study drug regimen will have a lower rate of puerperal infection than the placebo group.

Nulliparous women with obesity who are undergoing induction of labor at term will be eligible for participation in the study. Across all sites, 787 total subjects will be recruited.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥30
* No prior deliveries at or beyond 20 weeks gestation
* Undergoing induction of labor
* Gestational age 37 weeks or more
* Age 15-45
* Not receiving IAP for GBS prophylaxis

Exclusion Criteria:

* Fetal death prior to labor induction
* Known fetal anomaly
* Multiple gestation
* Ruptured membranes for more than 12 hours
* Chorioamnionitis or other infection requiring antibiotics at the start of the labor induction
* Previous myometrial surgery
* Allergy to azithromycin or beta-lactam antibiotics

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — All subjects in this study will be pregnant women and fetus/infant dyads
Enrollment: 787 (Estimated)
Dates: Start 2025-04-29 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Rate of cesarean delivery | 30 days postpartum
  Determine whether a prophylactic antibiotic regimen during labor induction will decrease the rate of cesarean delivery in obese, nulliparous women undergoing induction of labor

SECONDARY OUTCOMES:
Rate of chorioamnionitis development | 30 days postpartum
  Defined clinically by fever and maternal and fetal signs such as tachycardia and uterine tenderness
Rate of endometritis | 30 days postpartum
  Maternal development of endometritis
Rate of cesarean wound infection | 30 days postpartum
  Rate of maternal would infection from cesarean section
Rate of postpartum hemorrhage | 30 days postpartum
  Rate of maternal postpartum hemorrhage
Rate of blood transfusion | 30 days postpartum
  Rate of maternal blood transfusions
Rate of intensive care unit admission | 30 days postpartum
  Maternal admission into intensive care unit
Rate of hospital readmission | 30 days postpartum
  Maternal hospital readmission after delivery
Rate of indications for cesarean delivery | 30 days postpartum
  Rate of indications for a cesarean delivery
Maternal hospital stay | 30 days postpartum
  Length of maternal hospital stay
Neonate hospital stay | 30 days postpartum
  Length of neonatal hospital stay
Rate of NICU admission | 30 days postpartum
  Neonatal intensive care unit (NICU) admission
APGAR score | 30 days postpartum
  5-minute APGAR score <4 (neonate)
Rate of respiratory distress syndrome | 30 days postpartum
  Development of infant respiratory distress syndrome
Rate of sepsis | 30 days postpartum
  Infant sepsis (either suspected or confirmed)
Rate of necrotizing enterocolitis | 30 days postpartum
  Infant necrotizing enterocolitis
Periventricular leukomalacia | 30 days postpartum
  Development of periventricular leukomalacia in infant as seen by ultrasound
Rate of intraventricular hemorrhage | 30 days postpartum
  Intraventricular hemorrhage grade III or higher
Neonatal death | 30 days postpartum
  Death of neonate

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Pierce, MD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No